CLINICAL TRIAL: NCT03901651
Title: Combined Forward and Retroflexion Withdrawal in the Detection of Polyps and Adenoma During Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RV03-2019
Record Dates: First submitted 2019-03-25; First posted 2019-04-03 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-06

CONDITIONS: Colonic Polyp; Colonic Neoplasms; Colonic Adenoma
Keywords: colonic polyps
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: Patients submitted for screening, surveillance or diagnostic colonoscopy. First, a colonoscopy using a HD standard colonoscope using a forward viewing withdrawal technique. Then, a second colonoscopy using the Retroview colonoscope combining forward and retroflexed evaluation of the colon will be performed in the same patient.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard colonoscopy (Active Comparator): Patients submitted for screening, surveillance or diagnostic colonoscopy. A standard colonoscopy with forwarding viewing withdrawal technique. An HD colonoscope with I-scan technology will be used by one expert endoscopist.
  Each polyp and adenoma will be recorded, including the size and location. Polyps will be removed before the second procedure.
  Interventions: Diagnostic Test: Colonoscopy with standard colonoscope and forward withdrawal technique
- Retroview colonoscopy (Experimental): The same group of patients. A second colonoscopy using a combined forward and retroflexed evaluation of the colonic mucosa. using the Retroview™ scope. The operator will be blind to the first colonoscopy findings.
  The operator will record the polyps and adenoma encountered, describing the size and location.
  Interventions: Diagnostic Test: Colonoscopy with Retroview scope combing forward and retroflexed withdrawal technique

INTERVENTIONS:
Diagnostic Test: Colonoscopy with Retroview scope combing forward and retroflexed withdrawal technique — Colonoscopy using a combined forward and retroflexed evaluation of the colonic mucosa. using the Retroview™ scope. The operator will be blind to the standard colonoscopy findings.
  The operator will record the polyps and adenoma encountered, describing the size and location.
  Arms: Retroview colonoscopy
Diagnostic Test: Colonoscopy with standard colonoscope and forward withdrawal technique — A standard colonoscopy with forwarding viewing withdrawal technique. An HD colonoscope with I-scan technology will be used by one expert endoscopist.
  Each polyp and adenoma will be recorded, including the size and location.
  Arms: Standard colonoscopy

SUMMARY:
Colonoscopy is the standard of care for the detection of colorectal polyps and adenoma, and colorectal cancer detection. Despite a meticulous evaluation of the colonic mucosa during colonoscopy, a substantial number of colorectal polyps might be missed and colorectal cancer might not be prevented.

Previous studies described a 12-28% of miss-rate for all polyps, a 31% for hyperplastic polyps and 6-27% for adenomas, with a higher miss rate noted for smaller polyps. The lesion missing rate depends on several factors, such as the location on difficult areas to be evaluated with conventional colonoscopes (the proximal side of the ileocecal valve, haustral folds, flexures or rectal valves), a flat shape, an inadequate bowel preparation and inadequate endoscopy technique, a time-limited colonoscope withdrawal.

If the standard 140º angle of view colonoscope is used approximately 13% of the colonic surface is unevaluated. The incorporation of colonoscopes with a 170-degree wide angled could improve adenoma detection rate.

The introduction of high definition (HD) colonoscopes and visual image enhancement technologies, such as narrow band imaging (NBI, Olympus America, Center Valley, PA), I-SCAN™ (Pentax Medical, Montvale, NJ) and Fuji Intelligent Chromo-Endoscopy (FICE™, Fujinon Endoscopy, Wayne, NJ) have improved the lesion characterization; however, several studies have failed to prove an increase in the adenoma detection rates.

The Third Eye Retroscope (Avantis Medical Systems, Sunnyvale, CA) is a disposable retrograde viewing device advanced through the accessory channel of a standard colonoscope. It allows retrograde viewing behind colonic folds and flexures simultaneously with the forward view of the colon. Although it shows an increase in the adenoma detection rate by 11%-25%, it has many disadvantages. First, it requires a separate processor and the device is disposable, increasing the cost of the procedure. Second, it occupies the working channel of the colonoscope, limiting the ability to suction. Third, if a polyp is detected, the viewing device has to be removed in order to perform the polypectomy. Fourth, the optic is not high definition and finally, the endoscopist has to get used to visualizing and processing two simultaneous video streams from the colonoscopy and from the retroscope device.

DETAILED DESCRIPTION:
The Retroview™ (Pentax Medical, HOYA Co.) colonoscope has a short turning radius at the colonoscope tip, that allows a retroflexed view of the colon during withdrawal. This might allow the detection of polyps hidden behind flexures, folds, and valves, from the cecum to the rectum.

This device offers many advantages, such as the ability to provide a high definition view of the proximal aspects of colonic folds, flexures, and valves with no additional equipment or device costs. The image quality is high definition and the colonoscope also incorporates the I-SCAN technology. The suction/work channel of the colonoscope is available for therapeutic procedures. Polypectomy can be performed with the colonoscope during retroflexion, without losing view of the polyp. The only disadvantages are the higher consumed withdrawal time because the additional retroflexed withdrawal to the standard withdrawal and that a small portion of the colon is obscured by the shaft of the colonoscope in retroflexion that may be the reason why combined standard withdrawal with retroflexed withdrawal has proved to be better than retroflexed withdrawal alone.

The aim of this study is to determinate the polyp and adenoma detection rate via performing a colonoscopy using a conventional scope with standard withdrawal (forward view) and a combined forward and retroflexed withdrawal technique using the RetroView™ colonoscope.

Lesion's dimensions and characteristics will be recorded to determine a difference between both techniques.

MATERIALS AND METHODS Setting: Instituto Ecuatoriano de Enfermedades Digestivas (IECED), Omni Hospital Academic Tertiary Center. We will include patients from January 2019 to November 2019. The study protocol and consent form has been approved by the Institutional Review Board of our institution and will be conducted according to the Declaration of Helsinki. Patients will provide written informed consent.

Intervention: endoscopic technique. Participants will be submitted to two colonoscopies on the same day. First, a standard colonoscopy will be performed using a conventional HD colonoscope with I-Scan (EC 3490LK, PENTAX, Montvale, NJ) that has a 13.2 mm tube diameter and a total length of 2023 mm). Then a second procedure, combining the standard forward view and retroflexed withdrawal will be performed using the Retroview™ colonoscope (EC34-i10TL, Pentax Medical, Montvale, NJ), that has an 11.6 mm tube diameter and 2023 mm length.

The endoscopy images will be seen on a 27-inch, flat panel, HD LCD monitor (Radiance™ ultra-SC-WU27-G1520 model). All participants will have the same colonic preparation with 4 liters of polyethylene glycol (PEG) the day before and bowel preparation will be evaluated using the Boston Bowel Preparation Scale.

Two endoscopists with proficiency in retroflexed withdrawal will perform the colonoscopies. Colonoscopies will be performed in a tandem, random manner. First one endoscopist will perform the conventional colonoscopy using standard withdrawal technique with standard colonoscopes and then the second endoscopist blinded to the first colonoscopy results will perform the second colonoscopy with the Retroview scope and combination withdrawal (retroflexed with standard withdrawal). The operator assigned to each colonoscopy will be chosen randomly. A minimum withdrawal time of 10 minutes will be required for each procedure. After the examination, endoscopist will fill a questionnaire describing each polyp and adenoma found, including the size and location. The withdrawal time spent in each procedure will be measured.

Statistical analysis: Baseline characteristics will be analyzed using Chi-square o Fisher Test for categorical variable and Mann-Whitney Test for continuous variables. If there is more than one polyp in one patient it will be considered individually for statistical purposes. A P value of less than 0.05 will be considered statistically significant. All the statistical analysis will be performed using R.

Limitations: The protocol will be performed in a single-center by six endoscopists. A lack of a control group because the intention is to compare two endoscopic techniques in the same setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients capable of providing written consent
* Colonoscopy indicated for colorectal cancer screening or surveillance
* Patients submitted for polypectomy
* Colonoscopy indicated for diagnostic purposes: anemia, abdominal pain, constipation, alteration of bowel habits.

Exclusion Criteria:

* Patients under 45 years and over 80 years of age.
* Pregnancy and/or nursing.
* Patients with past-medical history of cardiac, renal, hepatic or severe metabolic diseases
* Unable to tolerate sedation
* Severe uncontrolled coagulopathy
* Past surgical history of colonic resection, ileostomy or colostomy.
* Previous abdominal or pelvic radiation therapy.
* Patients with inflammatory bowel disease, polyposis syndrome or acute diverticulitis.
* Patients with high suspicion of colonic obstruction or history of prior obstruction.
* Patients with gastrointestinal bleeding.
* Inadequate bowel preparation. The bowel preparation will be evaluated using the Boston Bowel Preparation Scale. Patients with < 2 points in at least one of the three segments of the colon will be excluded.
* Patients who after the beginning of the colonoscopy have to be suspended due to the inability to reach into the cecum because of unfavorable anatomy or impassable tumors/stenosis.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Polyp detection rate with standard colonoscope and the Retroview colonoscope | 23 months
  Polyps found during standard colonoscopy/total of polyps found x 100; polyps found with the Retroview scope/total of polyps found x100. The total of polyps found will be defined by the combination of both methods
Adenoma detection rate with standard colonoscope and retroview colonoscope. | 23 months
  Adenomas found during standard colonoscopy/total of adenomas found x 100; adenomas found with the Retroview scope/total of adenomas found x100. The total of adenomas found will be defined by the combination of both methods

SECONDARY OUTCOMES:
Lesion miss rate with the standard colonoscope and Retroview scope | 23 months
  Lesion miss rate: missed lesions/ total of lesions (polyps and adenomas) x100
Number of lesions (adenomas and polyps) detected with the standard colonoscope and Retroview colonoscope. | 23 months
  The number of lesions will be described in each patient from both procedures.
Size of lesions (adenomas and polyps) detected with the standard colonoscope and Retroview colonoscope. | 23 months
  The size of lesions (adenomas and polyps) detected with the standard colonoscope and Retroview colonoscope. The size will be measured using a standard biopsy forceps as a comparison method.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, MC, Principal Investigator — Instituto Ecuatoriano de Enfermedades Digestivas
Locations (1):
- Ecuadorian Institute of Digestive Diseases, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No